CLINICAL TRIAL: NCT02518815
Title: Preoperative Active Warming Prevents Postoperative Hypothermia in Patients Undergoing Laparoscopic Gynecologic Surgery. A Randomized Control Trial
Brief Title: Preoperative Warming Prevents Postoperative Hypothermia in Laparoscopic Gynecologic Surgery. A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Garron Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 550-1304-Mis-213
Record Dates: First submitted 2015-07-22; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Hypothermia Following Anesthesia; Hypothermia; Hypothermia, Accidental; Body Temperature Changes; Hypothermia Due to Anesthetic
MeSH Terms: conditions — Hypothermia; Body Temperature Changes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prewarming group (Experimental): Prewarmed for 20 minutes prior to OR using 3M Bair Paws System, a forced air warming blanket. This warming blanket was then used intraoperatively throughout the case.
  Interventions: Device: 3M Bair Paws Warming System
- Control group (No Intervention): Patients received standard care, which is no active prewarming prior to OR. A full body, forced air warming blanket (same as treatment group) was used intraoperatively throughout the case.

INTERVENTIONS:
Device: 3M Bair Paws Warming System — 20 minutes of prewarming immediately pre-operatively using 3M Bair Paws warming system
  Arms: Prewarming group

SUMMARY:
This study examined whether 20 minutes of prewarming prior to gynecological laparoscopic surgery prevented inadvertent post-operative hypothermia. Treatment group received prewarming using a forced air body warming, control group received no active warming system. Both groups were then warmed with forced air warmer intraoperatively.

DETAILED DESCRIPTION:
Inadvertent perioperative hypothermia is a well known perioperative complication. The behavioural response to hypothermia is the most powerful protective tool, more effective than any autonomic response, and is obviously removed in the operative setting. Anesthesia alters thermoregulation by profoundly changing the thresholds for vasoconstriction and shivering, making patients vulnerable to the adverse outcomes related to mild hypothermia. Inadvertent postoperative hypothermia can occur in up to 70% of surgical patients. It is defined as a core temperature below 36°C (96.8°F). The aim of this study was to determine if prewarming with an active warming system for 20 minutes preoperatively could prevent postoperative inadvertent hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* undergoing elective laparoscopic gynecological surgical procedures
* expected duration >60 minutes
* BMI 18-45

Exclusion Criteria:

* Current fever (temperature>38.1°C)
* active endocrine disorders were exclusion criteria

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Oral temperature immediately postoperatively | Immediately post-operatively
  Immediate postoperative oral temperature on admission to the post-anesthetic care unit.

SECONDARY OUTCOMES:
Oral temperature 30 minutes postoperatively | 30 min after admission to post-anesthetic care unit
  Oral temperature 30 minutes after admission to the post-anesthetic care unit.
Oral temperature at discharge from post-anesthetic care unit | Discharge from post-anesthetic care unit (average 99 minutes)
  Oral temperature upon discharge from the post-anesthetic care unit.
11-point Pain score | 30 min after admission to post-anesthetic care unit
  11-point VAS pain score postoperatively measured 30 minutes after admission to the post-anesthetic care unit

CONTACTS AND LOCATIONS:
Overall Officials: James Kulchyk, MD, Principal Investigator — Michael Garron Hospital
Locations (1):
- Toronto East General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Bellamy C. Inadvertent hypothermia in the operating theatre: an examination. J Perioper Pract. 2007 Jan;17(1):18-25. doi: 10.1177/175045890701700102. PMID 17265749
- [Background] Kurz A. Physiology of thermoregulation. Best Pract Res Clin Anaesthesiol. 2008 Dec;22(4):627-44. doi: 10.1016/j.bpa.2008.06.004. PMID 19137807
- [Background] Annadata R, Sessler DI, Tayefeh F, Kurz A, Dechert M. Desflurane slightly increases the sweating threshold but produces marked, nonlinear decreases in the vasoconstriction and shivering thresholds. Anesthesiology. 1995 Dec;83(6):1205-11. doi: 10.1097/00000542-199512000-00011. PMID 8533913
- [Background] Kurz A, Go JC, Sessler DI, Kaer K, Larson MD, Bjorksten AR. Alfentanil slightly increases the sweating threshold and markedly reduces the vasoconstriction and shivering thresholds. Anesthesiology. 1995 Aug;83(2):293-9. doi: 10.1097/00000542-199508000-00009. PMID 7631951
- [Background] Matsukawa T, Kurz A, Sessler DI, Bjorksten AR, Merrifield B, Cheng C. Propofol linearly reduces the vasoconstriction and shivering thresholds. Anesthesiology. 1995 May;82(5):1169-80. doi: 10.1097/00000542-199505000-00012. PMID 7741292
- [Background] Talke P, Tayefeh F, Sessler DI, Jeffrey R, Noursalehi M, Richardson C. Dexmedetomidine does not alter the sweating threshold, but comparably and linearly decreases the vasoconstriction and shivering thresholds. Anesthesiology. 1997 Oct;87(4):835-41. doi: 10.1097/00000542-199710000-00017. PMID 9357885
- [Background] Sessler DI. Perioperative thermoregulation and heat balance. Ann N Y Acad Sci. 1997 Mar 15;813:757-77. doi: 10.1111/j.1749-6632.1997.tb51779.x. PMID 9100967
- [Background] Buggy DJ, Crossley AW. Thermoregulation, mild perioperative hypothermia and postanaesthetic shivering. Br J Anaesth. 2000 May;84(5):615-28. doi: 10.1093/bja/84.5.615. No abstract available. PMID 10844839
- [Background] Doufas AG. Consequences of inadvertent perioperative hypothermia. Best Pract Res Clin Anaesthesiol. 2003 Dec;17(4):535-49. doi: 10.1016/s1521-6896(03)00052-1. PMID 14661656
- [Background] Reynolds L, Beckmann J, Kurz A. Perioperative complications of hypothermia. Best Pract Res Clin Anaesthesiol. 2008 Dec;22(4):645-57. doi: 10.1016/j.bpa.2008.07.005. PMID 19137808
- [Background] Kurz A, Sessler DI, Lenhardt R. Perioperative normothermia to reduce the incidence of surgical-wound infection and shorten hospitalization. Study of Wound Infection and Temperature Group. N Engl J Med. 1996 May 9;334(19):1209-15. doi: 10.1056/NEJM199605093341901. PMID 8606715
- [Background] Sessler DI, Schroeder M, Merrifield B, Matsukawa T, Cheng C. Optimal duration and temperature of prewarming. Anesthesiology. 1995 Mar;82(3):674-81. doi: 10.1097/00000542-199503000-00009. PMID 7879936
- [Background] Vanni SM, Braz JR, Modolo NS, Amorim RB, Rodrigues GR Jr. Preoperative combined with intraoperative skin-surface warming avoids hypothermia caused by general anesthesia and surgery. J Clin Anesth. 2003 Mar;15(2):119-25. doi: 10.1016/s0952-8180(02)00512-3. PMID 12719051
- [Background] Hocker J, Bein B, Bohm R, Steinfath M, Scholz J, Horn EP. Correlation, accuracy, precision and practicability of perioperative measurement of sublingual temperature in comparison with tympanic membrane temperature in awake and anaesthetised patients. Eur J Anaesthesiol. 2012 Feb;29(2):70-4. doi: 10.1097/EJA.0b013e32834cd6de. PMID 22037543
- [Background] Amoateng-Adjepong Y, Del Mundo J, Manthous CA. Accuracy of an infrared tympanic thermometer. Chest. 1999 Apr;115(4):1002-5. doi: 10.1378/chest.115.4.1002. PMID 10208200
- [Background] Frank SM, Fleisher LA, Breslow MJ, Higgins MS, Olson KF, Kelly S, Beattie C. Perioperative maintenance of normothermia reduces the incidence of morbid cardiac events. A randomized clinical trial. JAMA. 1997 Apr 9;277(14):1127-34. PMID 9087467
- [Background] Melling AC, Ali B, Scott EM, Leaper DJ. Effects of preoperative warming on the incidence of wound infection after clean surgery: a randomised controlled trial. Lancet. 2001 Sep 15;358(9285):876-80. doi: 10.1016/S0140-6736(01)06071-8. PMID 11567703
- [Background] Schmied H, Kurz A, Sessler DI, Kozek S, Reiter A. Mild hypothermia increases blood loss and transfusion requirements during total hip arthroplasty. Lancet. 1996 Feb 3;347(8997):289-92. doi: 10.1016/s0140-6736(96)90466-3. PMID 8569362
- [Background] Winkler M, Akca O, Birkenberg B, Hetz H, Scheck T, Arkilic CF, Kabon B, Marker E, Grubl A, Czepan R, Greher M, Goll V, Gottsauner-Wolf F, Kurz A, Sessler DI. Aggressive warming reduces blood loss during hip arthroplasty. Anesth Analg. 2000 Oct;91(4):978-84. doi: 10.1097/00000539-200010000-00039. PMID 11004060
- [Background] Horn EP, Bein B, Bohm R, Steinfath M, Sahili N, Hocker J. The effect of short time periods of pre-operative warming in the prevention of peri-operative hypothermia. Anaesthesia. 2012 Jun;67(6):612-7. doi: 10.1111/j.1365-2044.2012.07073.x. Epub 2012 Feb 29. PMID 22376088
- [Background] Ott DE, Reich H, Love B, McCorvey R, Toledo A, Liu CY, Syed R, Kumar K. Reduction of laparoscopic-induced hypothermia, postoperative pain and recovery room length of stay by pre-conditioning gas with the Insuflow device: a prospective randomized controlled multi-center study. JSLS. 1998 Oct-Dec;2(4):321-9. PMID 10036122
- [Background] Makinen MT. Comparison of body temperature changes during laparoscopic and open cholecystectomy. Acta Anaesthesiol Scand. 1997 Jun;41(6):736-40. doi: 10.1111/j.1399-6576.1997.tb04775.x. PMID 9241334
- [Background] Luck AJ, Moyes D, Maddern GJ, Hewett PJ. Core temperature changes during open and laparoscopic colorectal surgery. Surg Endosc. 1999 May;13(5):480-3. doi: 10.1007/s004649901017. PMID 10227947
- [Background] Peng Y, Zheng M, Ye Q, Chen X, Yu B, Liu B. Heated and humidified CO2 prevents hypothermia, peritoneal injury, and intra-abdominal adhesions during prolonged laparoscopic insufflations. J Surg Res. 2009 Jan;151(1):40-7. doi: 10.1016/j.jss.2008.03.039. Epub 2008 Apr 23. PMID 18639246
- [Background] Nelskyla K, Yli-Hankala A, Sjoberg J, Korhonen I, Korttila K. Warming of insufflation gas during laparoscopic hysterectomy: effect on body temperature and the autonomic nervous system. Acta Anaesthesiol Scand. 1999 Nov;43(10):974-8. doi: 10.1034/j.1399-6576.1999.431002.x. PMID 10593458
- [Background] Fernandes LA, Braz LG, Koga FA, Kakuda CM, Modolo NS, de Carvalho LR, Vianna PT, Braz JR. Comparison of peri-operative core temperature in obese and non-obese patients. Anaesthesia. 2012 Dec;67(12):1364-9. doi: 10.1111/anae.12002.x. Epub 2012 Oct 22. PMID 23088746
- [Background] Nguyen NT, Fleming NW, Singh A, Lee SJ, Goldman CD, Wolfe BM. Evaluation of core temperature during laparoscopic and open gastric bypass. Obes Surg. 2001 Oct;11(5):570-5. doi: 10.1381/09608920160557039. PMID 11594097
- [Background] De Witte JL, Demeyer C, Vandemaele E. Resistive-heating or forced-air warming for the prevention of redistribution hypothermia. Anesth Analg. 2010 Mar 1;110(3):829-33. doi: 10.1213/ANE.0b013e3181cb3ebf. Epub 2009 Dec 30. PMID 20042439